CLINICAL TRIAL: NCT03358862
Title: Myopia Progression in Children and Adolescents Before and After Use of a Novel Extended Depth of Focus Daily Disposable Soft Contact Lens
Brief Title: Myopia Progression With a Novel Extended Depth of Focus Contact Lens
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aller, Thomas A., OD (Other)
Collaborators: Visioneering Technologies, Inc (Industry)
Responsible Party: Principal Investigator, Thomas A. Aller, OD, Principal Investigator, Aller, Thomas A., OD
Other Study IDs: SI-09-37
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Myopia; Myopia, Progressive
Keywords: myopia; progressive myopia; contact lenses; extended depth of focus; retrospective clinical series; axial length; refractive error
MeSH Terms: conditions — Myopia; Myopia, Degenerative; Refractive Errors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Myopes: Children, adolescents and young adults with existing progressive myopia equal to or exceeding -0.50 D in the year prior to beginning the use of the NaturalVue contact lens.
  Interventions: Device: NaturalVue Multifocal Contact Lens

INTERVENTIONS:
Device: NaturalVue Multifocal Contact Lens — NaturalVue multifocal contact lenses are daily disposable, distance center, multifocals with a novel extended depth of focus optical design. Patients wearing their habitual corrections who opt to change to this new lens will have their myopia progression monitored for up to two years.

SUMMARY:
Myopia has been increasing in prevalence and severity throughout the world over the last 30 years. Increasing levels of myopia are associated with increased frequencies and severity of various ocular pathologies, including cataracts, glaucoma, retinal detachments and other retinal pathologies and myopic maculopathy. Slowing myopia progression at a young age before the eye reaches excessive axial length may help to reduce the future risks of these ocular pathologies.

Conventional spectacles and contact lenses are prescribed correct myopia by moving the central focus of the eye for distance viewing from in front of the retina to on the retina centrally, or at the fovea. To varying degrees, these lenses allow the light to focus behind the retina, at varying peripheral retinal locations. These findings have led to efforts to design spectacle and contact lenses which correct peripheral hyperopic defocus, to reduce myopia progression.

The consensus theory for how both multifocal contact lenses and orthokeratology can control myopia progression is that they each can reduce, eliminate, or reverse relative peripheral hyperopic defocus. Existing published studies on the use of multifocal contact lenses to control myopia in humans have utilized lenses with the distance correction in the center with peripheral plus power to correct the peripheral blur. Until recently, there have been no daily disposable multifocal lenses in the US market with distance center designs.

The NaturalVue contact lens from Visioneering Technologies, Inc. is the first daily disposable distance center multifocal in the US. It has a novel extended depth of focus design where the distance correction is in the center of the optical zone, surrounded by a zone characterized by having a seamless, rapid transition from the distance power to a highly plus power at the edge of the optical zone.

This study will analyze the myopia progression of patients in the investigator's practice while wearing their habitual visual corrections for periods up to two years prior to being switched to NaturalVue contact lenses. They will then be followed for up to two years after beginning use of this novel lens design and the differences in their myopia progression after versus before this novel lens will be analyzed. Axial lengths will be measured with the IOLMaster after switching to NaturalVue, at six-month intervals and will be compared to axial lengths which have been collected with habitual corrections.

DETAILED DESCRIPTION:
Myopia has been increasing in prevalence and severity throughout the world over the last 30 years. Increasing levels of myopia are associated with increased frequencies and severity of various ocular pathologies, including cataracts, glaucoma, retinal detachments and other retinal pathologies and myopic maculopathy. Slowing myopia progression at a young age before the eye reaches excessive axial length may help to reduce the future risks of these ocular pathologies.

Conventional spectacles and contact lenses are prescribed to correct myopia by moving the central focus of the eye for distance viewing from in front of the retina to on the retina centrally, or at the fovea. To varying degrees, these lenses allow the light to focus behind the retina, at varying peripheral retinal locations. These findings have led to efforts to design spectacle and contact lenses which correct peripheral blur to reduce myopia progression.

The consensus theory for how both multifocal contact lenses and orthokeratology can control myopia progression is that they each can reduce, eliminate, or reverse relative peripheral hyperopic defocus. Existing published studies on the use of multifocal contact lenses to control myopia in humans have utilized lenses with the distance correction in the center with peripheral plus power to correct the peripheral hyperopic defocus. Until recently, there have been no daily disposable multifocal lenses in the US market with distance center designs.

The NaturalVue contact lens from Visioneering Technologies, Inc. is the first daily disposable distance center multifocal in the US. It has a novel extended depth of focus design where the distance correction is in the center of the optical zone, surrounded by a zone with a seamless, rapid transition from the distance power to a highly plus power at the edge of the optical zone.

This study will analyze the myopia progression of patients in the investigator's practice while wearing their habitual visual corrections for periods up to two years prior to being switched to NaturalVue contact lenses. They will then be followed for up to two years after beginning use of this novel lens design and the differences in their myopia progression after NaturalVue versus before NaturalVue will be analyzed. Axial lengths will be measured with the IOLMaster after switching to NaturalVue, at six-month intervals and will be compared to axial lengths which have been collected with habitual corrections.

ELIGIBILITY:
Inclusion Criteria:

* Myopic refractive error
* Astigmatism less than -2.50 D
* Evidence from clinical record of myopia progression equal to or greater than -0.50 D in at least one eye since the prior examination
* Ability to see 20/30 or better in the worse eye and 20/25 or better binocularly after one week adaptation
* Ability to properly insert, remove and care for study lens

Exclusion Criteria:

* Moderate to severe allergic conjunctivitis
* Moderate to severe dry eyes
* Keratoconus or other related corneal irregularity
* Strabismus
* Amblyopia
* Nystagmus

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population will be drawn from the clinic of the principal investigator.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Refractive error changes | Data will be collected at baseline and at every six months.
  Changes in myopia over time will be characterized by the spherical equivalent refractive error as measured by manifest subjective refraction.
Axial length of the eye | Data will be collected at baseline and at every six months.
  Changes in the axial length of the eye will be measured with the Zeiss IOLMaster

SECONDARY OUTCOMES:
Corneal curvature | Data will be collected at baseline and at every six months
  Keratometry will be measured by the Zeiss IOLMaster
Vitreous Chamber Depth | Data will be collected at baseline and at every six months.
  Vitreous Chamber Depth will be derived from measures of the Anterior Chamber Depth and the axial length as measured by the Zeiss IOLMaster.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Aller, OD, Principal Investigator — Independent
Locations (1):
- Dr. Thomas Aller Optometrist, Inc., San Bruno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aller TA, Liu M, Wildsoet CF. Myopia Control with Bifocal Contact Lenses: A Randomized Clinical Trial. Optom Vis Sci. 2016 Apr;93(4):344-52. doi: 10.1097/OPX.0000000000000808. PMID 26784710
- [Background] Aller TA. Clinical management of progressive myopia. Eye (Lond). 2014 Feb;28(2):147-53. doi: 10.1038/eye.2013.259. Epub 2013 Dec 20. PMID 24357844
- [Background] Aller TA, Wildsoet C. Bifocal soft contact lenses as a possible myopia control treatment: a case report involving identical twins. Clin Exp Optom. 2008 Jul;91(4):394-9. doi: 10.1111/j.1444-0938.2007.00230.x. PMID 18601670
- [Background] Cooper J, O'Connor B, Watanabe R, Fuerst R, Berger S, Eisenberg N, Dillehay SM. Case Series Analysis of Myopic Progression Control With a Unique Extended Depth of Focus Multifocal Contact Lens. Eye Contact Lens. 2018 Sep;44(5):e16-e24. doi: 10.1097/ICL.0000000000000440. PMID 29053555
- [Background] Woods J, Guthrie SE, Keir N, Dillehay S, Tyson M, Griffin R, Choh V, Fonn D, Jones L, Irving E. Inhibition of defocus-induced myopia in chickens. Invest Ophthalmol Vis Sci. 2013 Apr 12;54(4):2662-8. doi: 10.1167/iovs.12-10742. PMID 23471891